CLINICAL TRIAL: NCT03835403
Title: Public Access Defibrillation by Activated Citizen First-responders - The HeartRunner Trial
Brief Title: The HeartRunner Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Fredrik Folke, MD, PhD, Head of Research, Emergency Medical Services, Capital Region, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The HeartRunner Trial
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Usual Care (control arm) (No Intervention): These cardiac arrests will receive standard EMS response.
- HeartRunner Activation (Experimental): For these cardiac arrests, HeartRunners will be activated in addition to standard EMS response.
  Interventions: Other: Activation of HeartRunners

INTERVENTIONS:
Other: Activation of HeartRunners — Activation of volunteer citizen first-responders to respond to nearby cardiac arrests
  Arms: HeartRunner Activation

SUMMARY:
The study will assess 30-day survival for cases where volunteer citizen responders ('heart runners') were activated through a smartphone app to retrieve an AED in case of suspected out-of-hospital cardiac arrest (OHCA) versus standard emergency medical services care. The study will randomize emergency medical dispatch center incoming calls which are suspected out-of-hospital cardiac arrest, such that half will be randomized to activation of heart runners and half to no activation of heart runners (standard care). The study will also assess physical or psychological risks involved for the activated heart runners.

DETAILED DESCRIPTION:
Chances of survival after out-of-hospital cardiac arrest decrease 10% per minute from collapse until defibrillation. Activating volunteer citizens through the emergency medical dispatch center can potentially increase rates of bystander defibrillation and survival. The HeartRunner trial will investigage the effect of activating registered volunteer citizens through a mobile app integrated with the emergency medical services on 30-day survival following out-of-hospital cardiac arrest. Both arms will receive standard care by the Emergency Medical Services. The intervention arm will additionally receive the activation of volunteer citizen responders. The randomization will take place independently in 3 different strata according to heart runner distance to OHCA (< 3 min, 3-9 min, > 9 min). The trial will also assess whether it is safe, both physically and psychologically, to activate volunteer citizen responders to respond to out-of-hospital cardiac arrests.

ELIGIBILITY:
Inclusion Criteria:

* All out-of-hospital cardiac arrests recognized by Emergency Medical Dispatcher and where the HeartRunner system is activated.
* Non-traumatic etiology, this excludes intoxication, drowning or suicide.
* Age > 7 years

Exclusion Criteria:

* Caller is not in direct contact with the patient
* If Emergency Medical Dispatcher deems AED is not indicated, e.g., in nursing homes where trained personal is present.
* OHCAs not treated by the EMS due to ethical reasons or obvious signs of death
* OHCAs with no heart runners within 1800 meters
* Not true cardiac arrest (suspected, but not verified)
* EMS-witnessed OHCAs

Emergency medical dispatchers are instructed not to activate heart runners in case any of the exclusion criteria above. However, since it can be challenging for emergency medical dispatchers to gather sufficient information about the patient within the first few minutes, heart runners will admittedly be activated even though they should not have been. Since randomization will occur for all cases in which a heart runner is activated, cases with any of the exclusion criteria will be secondarily excluded.

These cases will be accounted for but not included in analyses of outcome. Our pilot study showed approximately 60% of suspected cardiac arrests were true cardiac arrests. Therefore, we expect 40% of cases for which heart runners were dispatched not to be true cardiac arrests.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
30-day survival | 30 days after date of out-of-hospital cardiac arrest
  Patient alive 30 days after date of out-of-hospital cardiac arrest

SECONDARY OUTCOMES:
Rates of bystander defibrillation | During cardiac arrest
  Percentage of patients who received defibrillation prior to EMS arrival
Rates of bystander cardiopulmonary resuscitation | During cardiac arrest
  Percentage of patients who received bystander cardiopulmonary resuscitation prior to EMS arrival
Rates of return of spontaneuous circulation | Immediately after out-of-hospital cardiac arrest
  sustained circulation indicating successful resuscitation
Rates of survival after 1 year | 1 year after date of out-of-hospital cardiac arrest
  percentage of patients alive 1 year after out-of-hospital cardiac arrest
Rates of neurological intact survival | At hospital discharge
  percentage of patients with cerebral performance category score of 1-2

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Folke, MD, PhD, Principal Investigator — Copenhagen EMS
Locations (1):
- Emergency Medical Services Copenhagen, Copenhagen, Ballerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mottlau KH, Andelius LC, Gregersen R, Malta Hansen C, Folke F. Citizen Responder Activation in Out-of-Hospital Cardiac Arrest by Time of Day and Day of Week. J Am Heart Assoc. 2022 Feb;11(3):e023413. doi: 10.1161/JAHA.121.023413. Epub 2022 Jan 21. PMID 35060395
- [Derived] Andelius L, Malta Hansen C, Lippert FK, Karlsson L, Torp-Pedersen C, Kjaer Ersboll A, Kober L, Collatz Christensen H, Blomberg SN, Gislason GH, Folke F. Smartphone Activation of Citizen Responders to Facilitate Defibrillation in Out-of-Hospital Cardiac Arrest. J Am Coll Cardiol. 2020 Jul 7;76(1):43-53. doi: 10.1016/j.jacc.2020.04.073. PMID 32616162

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Updated protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03835403/Prot_SAP_002.pdf
  • Study Protocol: Changes to protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03835403/Prot_004.pdf
  • Statistical Analysis Plan: Detailed Final Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03835403/SAP_003.pdf